CLINICAL TRIAL: NCT04253886
Title: Comparison of the Fekry Oral Intubating Airway and Ovassapian Fibreoptic Intubating Airway for Fibreoptic Orotracheal Intubation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: N 31-2018/Ms
Record Dates: First submitted 2020-01-21; First posted 2020-02-05 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Ovassapian VS Fekry Airways

STUDY DESIGN:
Intervention Model Description: Either the Fekry Oral Airway Intubator (Ameco Tech, Cairo, Egypt) or the Ovassapian Fibreoptic Intubating Airway (Kendall Sheridan, Argyle, NY) will be inserted into the mouth in random order, and the patient's lungs ventilated by bag and facemask with 100% oxygen and 1-1.5% isoflurane. Blinding will be impossible in this study as the operator has to see the airway through the fibrescope in order to perform the assessment.
  After confirmation of full neuromuscular blockade, a bronchoscope with a preloaded tracheal tube will be then inserted through the airway for bronchoscopic assessment.
Who Masked: Participant, Investigator
Masking Description: Randomization will be done using computer generated number and concealed using sequentially numbered, sealed opaque envelope.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): The Ovassapian Fibreoptic Intubating Airway has a flat lingual surface that widens distally. This provides better retraction of the tongue to prevent it and the soft tissues of the anterior pharyngeal wall from herniating around the side of the airway. The airway has a pair of vertical sidewalls and two pairs of curved guide walls at its proximal section. These walls are separated by a gap which allows removal of the airway after intubation has been completed
  Interventions: Device: Ovassapian Fibreoptic Intubating Airway
- Group B (Active Comparator): Fekry airway:
  ● It has two parts are: Airway body& Special connector
  1. Airway body consists of:
     1. Flange → it is the buccal end it is 7 cm wide to prevent it from
     2. moving deeper into mouth & may also serve to fix airway in place.
     3. Bite Portion → it is straight & fits between teeth &oral cavity.
     4. Oral straight part → open anterior lingual part; it varies in length according to size
     5. Pharyngeal curved part → extends backwards to correspond the shape oropharynx and ends below laryngeal inlet.
  2. The connector: it is a special type (two sizes: adult and pediatric) can attach to all ventilating machines& it has a teeth rest act as a bite block.
  Interventions: Device: Ovassapian Fibreoptic Intubating Airway

INTERVENTIONS:
Device: Ovassapian Fibreoptic Intubating Airway — The fibreoptic bronchoscope remains one of the most important methods of intubating patients particularly when there is difficulty with intubation.Facilitating fiberoptic oropharyngeal intubation procedure, specific airways have been devised to push the tongue anteriorly to clear a passage for the fibrescope into the trachea. Of these airways Ovassapian Fibreoptic Intubating Airway (Kendall, Argyle, New York, New York, USA) and Fekry Oral Intubating Airway (Ameco Tech, Cairo, Egypt).
  Other Names: Fekry airway

SUMMARY:
The fibreoptic bronchoscope remains one of the most important methods of intubating patients particularly when there is difficulty with intubation Facilitating fiberoptic oropharyngeal intubation procedure, specific airways have been devised to push the tongue anteriorly to clear a passage for the fibrescope into the trachea.

Of these airways Ovassapian Fibreoptic Intubating Airway (Kendall, Argyle, New York, New York, USA) and Fekry Oral Intubating Airway (Ameco Tech, Cairo, Egypt).

DETAILED DESCRIPTION:
Ovassapian Fibreoptic Intubating Airway :

The Ovassapian Fibreoptic Intubating Airway has a flat lingual surface that widens distally. This provides better retraction of the tongue to prevent it and the soft tissues of the anterior pharyngeal wall from herniating around the side of the airway. The airway has a pair of vertical sidewalls and two pairs of curved guide walls at its proximal section. These walls are separated by a gap which allows removal of the airway after intubation has been completed.

Fekry airway:

● It has two parts are: Airway body& Special connector

1. Airway body consists of:

   1. Flange → it is the buccal end it is 7 cm wide to prevent it from moving deeper into mouth & may also serve to fix airway in place.
   2. Bite Portion → it is straight & fits between teeth &oral cavity.
   3. Oral straight part → open anterior lingual part; it varies in length according to size
   4. Pharyngeal curved part → extends backwards to correspond the shape oropharynx and ends below laryngeal inlet.
2. The connector: it is a special type (two sizes: adult and pediatric) can attach to all ventilating machines& it has a teeth rest act as a bite block.

ELIGIBILITY:
Inclusion Criteria:

1. ASA 1 to3,
2. Aged 18 to 60 years
3. Who presented for elective surgery requiring tracheal intubation

Exclusion Criteria:

1. All patients with a past history of difficult tracheal intubation
2. Patients with signs of possible difficult tracheal intubation (including modified Mallampati score 3 or 4
3. Limited mouth opening, thyromental distance < 4 cm, limited neck movement or upper airway disease

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 350 (Actual)
Dates: Start 2019-01-05 (Actual); Primary Completion 2019-10-15 (Actual); Study Completion 2019-11-09 (Actual)

PRIMARY OUTCOMES:
Time of intubation | Up to 24 hours
  Success rate of Time of intubation

SECONDARY OUTCOMES:
Advancing the endotracheal tube over the bronchoscope | Up to 24 hours
  Easiness of advancing the endotracheal tube over the bronchoscope
Percentage of success of endotracheal tube insertion | Up to 24 hours
  Percentage of success of endotracheal tube insertion from 1st trial in the shortest time
Removal of the bronchoscope | Up to 24 hours
  Easiness of removal of the bronchoscope after intubation.
Complications | Up to 24 hours
  Incidence of complications

CONTACTS AND LOCATIONS:
Overall Officials: Randa Badawi, M.D, Principal Investigator — Cairo University; Maha M Ismail Youssef, M.D, Principal Investigator — Cairo University; Sara Farouk Habib, M.D, Principal Investigator — Cairo University; Eman A Ahmed, M.Sc., Principal Investigator — Cairo University; Ahmed Abdalla Mohamed, M.D, Principal Investigator — Cairo University
Locations (1):
- Maha Mohamed Ismail Youssef, Cairo, Egypt